CLINICAL TRIAL: NCT04482439
Title: Evaluation of Quality of Vision and Visual Outcomes With Bilateral Implantation of the AcrySof® Vivity Intraocular Lens With a Target of Slight Myopia in the Non-dominant Eye
Brief Title: Evaluation of Vision After Vivity IOL Implantation With a Target of Slight Myopia in the Non-dominant Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newsom Eye & Laser Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TN-20-001
Record Dates: First submitted 2020-07-17; First posted 2020-07-22 (Actual); Results first posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-01

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: This study is a single-arm unmasked clinical evaluation study of binocular distance-corrected near (40 cm) visual acuity, when the non-dominant eye is targeted for slight myopia, after successful bilateral cataract surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Vivity mini-monovision (Experimental): Subjects will have bilateral Vivity IOL implanted, with a target of slight myopia in the non-dominant eye.
  Interventions: Device: Vivity Extended Depth of Focus intraocular lens (IOL)

INTERVENTIONS:
Device: Vivity Extended Depth of Focus intraocular lens (IOL) — Bilateral implantation of the Vivity lens after cataract surgery, with slight myopia planned in the non-dominant eye.

SUMMARY:
The objective is to assess binocular distance-corrected near (40 cm) visual acuity of patients after uneventful cataract surgery with bilateral implantation of the AcrySof® Vivity Intraocular lens (IOL) when the non-dominant eye is targeted for slight myopia.

DETAILED DESCRIPTION:
This study is a single-arm unmasked clinical evaluation study of binocular distance-corrected near (40 cm) visual acuity, when the non-dominant eye is targeted for slight myopia, after successful bilateral cataract surgery. Subjects will be assessed pre-operatively, operatively and at 1 day, 1 month and 3 months post-operatively. Clinical evaluations will include administration of a visual disturbance questionnaire (QUVID), patient-reported spectacle independence questionnaire (PRSIQ), and a satisfaction questionnaire (IOLSAT), as well as measurement of bilateral visual acuity and manifest refraction.

ELIGIBILITY:
Inclusion Criteria:

* • Presenting for uncomplicated bilateral cataract surgery and have an interest in spectacle independence using an EDF IOL

  * Meet the requirements for on-label implantation of the EDF IOL
  * Gender: Males and Females.
  * Age: 40 or older.
  * Willing and able to provide written informed consent for participation in the study.
  * Willing and able to comply with scheduled visits and other study procedures.
  * Have good ocular health, with no pathology that compromises visual acuity (outside of residual refractive error and cataract)
  * Have regular corneal astigmatism with a magnitude that can be treated with a non-toric IOL or toric IOL.
  * Have 20/32 (0.2 logMAR) or better potential acuity in both eyes

Exclusion Criteria:

* • Irregular astigmatism (e.g. keratoconus)

  * Corneal pathology (e.g. scar, dystrophy, pterygium, severe dry eye)
  * Monocular status (e.g. amblyopia)
  * Previous radial keratotomy, corneal refractive surgery or other corneal surgery (e.g. corneal transplant, DSAEK, lamellar keratoplasty)
  * Previous anterior or posterior chamber surgery (e.g., vitrectomy, laser iridotomy)
  * Diabetic retinopathy
  * Macular pathology (e.g. ARMD, ERM)
  * History of retinal detachment
  * Subjects who have an unstable acute or chronic disease or illness that would confound the results of this investigation (e.g., immunocompromised, connective tissue disease, clinically significant atopic disease, diabetes, and any other such disease or illness), that are known to affect postoperative visual acuity.
  * Participation in any investigational drug or device trial within the previous 30 days prior to the start date of this trial (or currently participating).

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Newsom, MD, Principal Investigator — Newsom Eye & Laser Center
Locations (1):
- Newsom Eye and Laser Center, Sebring, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Vivity Monovision Group: Eyes bilaterally implanted with Vivity IOL with non-dominant eye targeted for -0.75D of myopia.
Period: Overall Study
Arm/Group | Vivity Monovision Group
Started | 35
Completed | 33
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Unrelated illness | 1

BASELINE CHARACTERISTICS:
Population: All subject who completed their 3M visit.
Arm/Group | Vivity Monovision Group
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Binocular Near Visual Acuity
Description: binocular distance-corrected near (40 cm) visual acuity at 3 months postoperative.
Time Frame: 3 months postop
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Vivity Monovision Group
Number analyzed (Participants) | 33
logMAR | 0.14 (0.10)

2. Secondary Outcome: Prediction Accuracy
Description: Percentage of eyes with postoperative refractive accuracy within 0.5D of target
Time Frame: 3 months postop
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Vivity Monovision Group
Number analyzed (Participants) | 33
Number analyzed (Eyes) | 66
Eyes | 56

3. Secondary Outcome: Spectacle Independence
Description: Percent of all patients who never or rarely wear spectacles for distance, intermediate or near vision 3 months postop (based on the Patient-Reported Spectacle Independence Questionnaire - "a little of the time" or "none of the time")
Time Frame: 3 months postop
Population: All subjects who completed 3M PRSIQ questionnaire successfully
Measure: Count of Participants; unit: Participants
Arm/Group | Vivity Monovision Group
Number analyzed (Participants) | 32
Participants | 26

4. Secondary Outcome: Patient Spectacle Independence
Description: Patients reporting rarely or never needing glasses overall
Time Frame: 3 months postop
Measure: Count of Participants; unit: Participants
Arm/Group | Vivity Monovision Group
Number analyzed (Participants) | 33
Participants | 23

5. Secondary Outcome: Number of Participants Rating Frequency of Visual Disturbances as "Never" or "Rarely"
Description: This is the frequency of subjects responding, "Never" or "Rarely" to a question about the frequency of glare, halos and starbursts.
Time Frame: 3 months postop
Measure: Count of Participants; unit: Participants
Arm/Group | Vivity Monovision Group
Number analyzed (Participants) | 33
Participants
  Glare frequency "never" or 'rarely" | 19
  Halos frequency "never" or "rarely" | 18
  Starbursts frequency "never" or "rarely" | 13

6. Secondary Outcome: Manifest Refraction
Description: Manifest refraction (residual spherical equivalent refraction)
Time Frame: 3 months postop
Population: Each subject had 1 eye targeted for plano, and one eye targeted for myopia. So, each row includes 33 eyes of 33 subjects.
Measure: Mean (Standard Deviation); unit: diopters
Units Other Than Participants: Eyes
Arm/Group | Vivity Monovision Group
Number analyzed (Participants) | 33
Number analyzed (Eyes) | 66
diopters
  Eyes targeted for plano: number analyzed (Eyes) | 33
  Eyes targeted for plano | .01 (.31)
  Eyes targeted for myopia: number analyzed (Eyes) | 33
  Eyes targeted for myopia | -.74 (0.39)

7. Secondary Outcome: Residual Cylinder
Description: Residual refractive cylinder after surgery
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: diopters
Units Other Than Participants: Eyes
Arm/Group | Vivity Mini-monovision
Number analyzed (Participants) | 33
Number analyzed (Eyes) | 66
diopters | 0.42 (0.30)

8. Secondary Outcome: Uncorrected Distance Visual Acuity
Description: Bilateral uncorrected distance visual acuity
Time Frame: 3 months postop
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Vivity Monovision Group
Number analyzed (Participants) | 33
logMAR | 0.02 (0.09)

9. Secondary Outcome: Uncorrected Intermediate Visual Acuity
Description: Bilateral uncorrected visual acuity at 66 cm
Time Frame: 3 months postop
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Vivity Monovision Group
Number analyzed (Participants) | 33
logMAR | 0 (.07)

10. Secondary Outcome: Uncorrected Near Visual Acuity
Description: Bilateral uncorrected near visual acuity at 40 cm
Time Frame: 3 months postop
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Vivity Monovision Group
Number analyzed (Participants) | 33
logMAR | 0.12 (0.1)

11. Secondary Outcome: Corrected Distance Visual Acuity
Description: Bliateral corrected distance visual acuity
Time Frame: 3 months postop
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Vivity Monovision Group
Number analyzed (Participants) | 33
logMAR | 0.01 (0.08)

12. Secondary Outcome: Distance Corrected Intermediate Visual Acuity
Description: Bliateral distance corrected visual acuity at 66 cm
Time Frame: 3 months postop
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Vivity Monovision Group
Number analyzed (Participants) | 33
logMAR | 0.02 (0.06)

ADVERSE EVENTS:
Time Frame: Surgery to 3 months
Arm/Group | Vivity Monovision Group
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-02): https://cdn.clinicaltrials.gov/large-docs/39/NCT04482439/Prot_SAP_000.pdf